CLINICAL TRIAL: NCT03695016
Title: Advancement of Physical Activity Prescription in Clinical Practice
Brief Title: Activity Prescription in Clinical Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Bonny Rockette-Wagner, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO17120265
Record Dates: First submitted 2018-09-28; First posted 2018-10-03 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Physical Activity; Sedentary Lifestyle
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: 3 month wait-listed control trial in which participants are randomized to immediate intervention or intervention after 3 months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and their referring physician will be aware of participant randomization. Only the intervention coach, who will also notify the participants of their assignment will be aware of the assignments; other study staff and the investigator will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Intervention (Experimental): Participants will receive the ActiveGOALS 13 week, online self-directed intervention for increasing aerobic physical activity and decreasing time spent sitting. The intervention is based on social-cognitive theory models of behavior changes and utilizes barrier recognition, problem solving, and monitoring of behavior to initiate behavior change. They will also receive weekly feedback from a coach and be provided with online, paper, and wearable tracking devices. They will also be provided with links to tools that support physical activity.
  Interventions: Behavioral: ActiveGOALs
- Wait-listed Control (Other): This group will receive a monthly newsletter with general health advice during the wait period (3 months). After the three month follow-up visit/ collection of outcomes they will be offered the ActiveGOALS intervention in its entirety.
  Interventions: Behavioral: ActiveGOALs

INTERVENTIONS:
Behavioral: ActiveGOALs — 13 week, online self-directed intervention. Once weekly sessions are based on social-cognitive theory models of behavior changes. Coaches will provide weekly feedback . Behavior tracking tools will be provided. Links to tools that support physical activity will also be provided.

SUMMARY:
Most adults do not achieve the US aerobic physical activity (PA) guidelines (≥150 minutes/week of at least moderate intensity PA). Inadequate PA is considered a major risk factor for cardio-metabolic diseases and other poor health outcomes. Recommendations now endorse PA in reducing risk for certain diseases. Unfortunately, low PA levels are seldom identified and treated within clinical practice. This study will build on previous prevention efforts by focusing on the identifying and treating low PA levels in adults clinical care patients and referring them to an intervention that is feasible for delivery through clinical care.

DETAILED DESCRIPTION:
This study involves designing/ implementing a patient-centered, individually-focused physical activity (PA) intervention designed for integration into clinical care. We will recruit adult patients (aged 21-70; n=80) from the general internal medicine practice of a local health system who are not meeting the US aerobic activity goal of 150 minutes/ week of at least moderate intensity PA and who can safely increase PA without supervision. As low PA levels have been associated with numerous poor health outcomes, the primary intervention goal will be achievement of the US PA goal. A secondary goal will be to reduce sedentary behavior (SED), which is related to poor health outcomes (independent of PA achievement). Intervention materials will be developed using a patient/provider centered approach and delivered weekly over 3 months via an existing online platform with participants self-tracking behavior outcomes will be examined using a three month wait-listed control design in which all participants will eventually receive the intervention.

ELIGIBILITY:
Inclusion Criteria:

* not meeting the recommended levels of aerobic PA and have been identified by their primary care provider (PCP) as able to increase their PA without supervision.

Exclusion Criteria:

* Participated in a goal setting intervention for physical activity or a translation of the Diabetes Prevention Program within the last 2 years.
* Non-ambulatory or planning a procedure that will cause them to be non-ambulatory in the next 6 months
* Pregnant or planning a pregnancy in the next 6 months
* Need a way to access to the internet-based platform, at least a 6th grade reading level.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Aerobic activity | 10 days of recording at 0 and 3 months
  Objectively measured change in moderate-vigorous activity between 0 and 3 months using ActiGraph accelerometer
Change in Step counts | 10 days of recording at 0 and 3 months
  Objectively measured change in step counts between 0 and 3 months using ActiGraph accelerometer
Change in sedentary behavior | 10 days of recording at 0 and 3 months
  Objectively measured change in sedentary behavior between 0 and 3 months using ActiGraph accelerometer

SECONDARY OUTCOMES:
self-efficacy | pre-intervention and 3 and 6 months post-intervention
  questionnaire developed for this study, uses a 10 point scale.
Referring physician- usability of physicians report | 3 months post-intervention
  Physician satisfaction with study reports using questionnaire developed for this study. Several likert scale-based questions to determine satisfaction with different aspects of the report (design, readability, and aspects of usability).
Change in Aerobic Activity | 10 days of recording pre and post-intervention (3 and 6 months post)
  Change in objectively measured moderate-vigorous activity from ActiGraph accelerometer
Change in Step counts | 10 days of recording pre and post-intervention (3 and 6 months post)
  Change in objectively measured step counts from ActiGraph accelerometer
Change in Sedentary behavior | 10 days of recording pre and post-intervention (3 and 6 months post)
  Change in objectively measured sedentary behavior from ActiGraph accelerometer
Patient experience | 3 and 6 months post-intervention
  patient experience survey designed for this study with the help of patient partners to gather feedback from participants. Feedback will be used in the development of future interventions.
Health-related Quality of Life- PROMIS-29 score | pre-intervention and 3 and 6 months post-intervention
  Promis 29- Likert scale based questionnaire that determines quality of life in 7 areas of health with 4 questions in each area.
Participant cost | pre-intervention and 3 and 6 months post-intervention
  Cost survey questionnaire developed specifically for this study to determine health and personal monetary costs associated with participation in this study.
Perceived Health Score | pre-intervention and 3 and 6 months post-intervention
  EQ-VAX- Determines current perception of health on a 0-100 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Bonny Rockette-Wagner, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rockette-Wagner B, Fischer GS, Kriska AM, Conroy MB, Dunstan D, Roumpz C, McTigue KM. Efficacy of an Online Physical Activity Intervention Coordinated With Routine Clinical Care: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2020 Nov 3;9(11):e18891. doi: 10.2196/18891. PMID 33141103